CLINICAL TRIAL: NCT04352582
Title: COVID-19 and Vaccination Attitudes
Acronym: VACAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Zurich (Other); University of Lausanne (Other)
Responsible Party: Principal Investigator, Blanchard-Rohner Geraldine, Consultant, University Hospital, Geneva
Other Study IDs: VACAT
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Survey respondants
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
The investigators want to study how the exposure to the covid-19 pandemic affects attitudes towards science and vaccination, and how other general attitudes and values are affected.

DETAILED DESCRIPTION:
The investigators will carry out a survey in the UK, asking the same 3 questions on vaccination as in a past survey in late 2019 to the same previous respondents, supplementing this with further questions on covid-19 exposure and attitudes towards, among others, individualism-collectivism, health policy as well as trust in science and institutions.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers who participated in the November 2019 survey on vaccination will be contacted.

Exclusion Criteria:

* People who have not participated in the November 2019 survey
* People unwilling to participate again

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Representative sample of UK population
Sampling Method: Probability Sample
Enrollment: 1194 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
How vaccination and other attitudes are affected by COVID | Over last six months
  Survey

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Blanchard-Rohner, MD-PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Survey, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Replication data to be shared yet anonymized